CLINICAL TRIAL: NCT00144768
Title: A Multicenter, Multinational, Open-Label Study of Anti-Laronidase Antibody Formation and Urinary GAG Levels in Patients With Mucopolysaccharidosis I (MPS I) Being Treated With Aldurazyme® (Laronidase).
Brief Title: A Study Investigating the Relationship Between the Development of Laronidase Antibody and Urinary GAG (Glycosaminoglycan) Levels in Aldurazyme® Treated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALID02003
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2013-04

CONDITIONS: Mucopolysaccharidosis I; Hurler's Syndrome; Hurler-Scheie Syndrome; Scheie's Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: laronidase — dose of 0.58mg/kg body weight IV every week
  Other Names: Recombinant Human Alpha-L-Iduronidase, Aldurazyme®

SUMMARY:
The purpose of this study is to determine whether the development of antibodies to laronidase in patients with MPS I receiving Aldurazyme® impairs the clearance of GAG substrate.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of MPS I confirmed by measurable signs and symptoms and deficient α-L-iduronidase activity (<10% of the lower limit of normal).
* For a patients receiving Aldurazyme therapy prior to study entry: Have available as baseline data the results of urinary GAG levels and IgG antibody titers collected prior to the patient's first Aldurazyme infusion.
* Provide signed, written informed consent prior to any protocol-related procedures being performed. Consent of a legally authorized guardian(s) is (are) required for patients under 18 years.

Exclusion Criteria:

* Have previously received Aldurazyme without the collection of baseline samples as specified.
* Have a suspected hypersensitivity to Aldurazyme or a know hypersensitivity to components of infusion solution.
* Have received a Hematopoietic Stem Cell Transplantation, injection fibroblast therapy, or major organ transplant.
* Are receiving chronic immunosuppressant therapy.
* Have a medical condition, serious intercurrent illness, or other extenuating circumstances that may interfere with study compliance including all prescribed evaluations and follow-up activities.
* Are pregnant or lactating
* Have received investigational drug within 30 days prior to study enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Urinary GAG (glycosaminoglycans) | Up to 4 years
Immunogenicity Testing | Up to 4 years

SECONDARY OUTCOMES:
Safety | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Childrens Hospital Los Angeles, Los Angles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin